CLINICAL TRIAL: NCT01608685
Title: Interferon Gamma Release Assays Versus Tuberculin Skin Testing for the Detection of Latent Tuberculosis Infection in Renal Transplant Recipients
Brief Title: Interferon Gamma Release Assays (IGRA) Testing Versus Tuberculin Skin Test in Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Ligue Pulmonaire Genevoise (Other)
Responsible Party: Principal Investigator, Jean-Paul Janssens, Associate Professor, Ligue Pulmonaire Genevoise
Other Study IDs: KH-2010
Record Dates: First submitted 2011-07-05; First posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Latent Tuberculosis Infection
Keywords: Tuberculosis; Latent tuberculosis infection; Immunosuppression; Renal transplant recipient
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal transplant recipients: Inclusion criteria: All renal transplant recipients followed by the Division of Nephrology aged above 18 years, and having accepted study protocol after informed consent

SUMMARY:
Interferon gamma release assays (IGRA) have been shown to be more specific and sensitive for the detection of tuberculosis (latent or active infection) than the tuberculin skin test (TST) in immunocompetent individuals. However, very little data are available concerning the relative performance of IGRA and TST in immunosuppressed individuals from other causes than HIV.

The investigators hypothesize that IGRAs would be more sensitive and specific than the TST in a group of renal transplant recipients under chronic immunosuppressive treatment for detecting latent tuberculosis infection.

DETAILED DESCRIPTION:
In a recent study (Triverio PA et al. "Interferon-gamma release assays versus tuberculin skin testing for detection of latent tuberculosis in haemodialysis patients". Nephrol Dial Transplant 2009; 24: 1952-6), the investigators had compared 2 IGRAs (T-SPOT.TB and Quantiferon Gold) with the TST and shown that one IGRA was clearly more sensitive than the TST but that both tests had a very low sensitivity for detecting prior TB.

This study applies the same protocol to renal transplant recipients undergoing routine annual check-up visits: questionnaire with detailed collection of risk factors for latent tuberculosis infection (LTBI), history of prior contact with tuberculosis (TB), BCG (Bacille of Calmette and Guerin vaccine), prior TB or LTBI, treatment for TB or LTBI, analysis of chest X-ray for signs of prior TB, on-going treatment, level of immunosuppression (CD4 lymphocytes), simultaneous blood sampling for T-SPOT.TB and Quantiferon Gold, and tuberculin skin testing.

ELIGIBILITY:
Inclusion Criteria:

* prior renal transplantation;
* age > 18;
* stable clinical condition

Exclusion Criteria:

* hypersensitivity to tuberculin skin testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed by the Division of Nephrology after renal transplantation, and undergoing routine annual check-ups, in stable clinical condition, aged above 18
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Agreement between results of QuantiFERON-Gold-in-tube and probability of latent tuberculosis infection | Up to 3 years
  Agreement between probability of latent tuberculosis infection - established on the basis of a questionnaire and chest X-ray - and results of QuantiFERON-Gold-in-tube is computed
Agreement between results of T-SPOT.TB and probability of latent tuberculosis infection | Up to 3 years
  Agreement between probability of latent tuberculosis infection - established on the basis of a questionnaire and chest X-ray - and result of T-SPOT.TB is computed

SECONDARY OUTCOMES:
Agreement between results of IGRA tests and TST in renal transplant recipients | Up to 3 years
  Agreement between results of IGRA testing and between each IGRA test and TST will be determined by computing kappa values

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hadaya, MD, Principal Investigator — Division of Nephrology/Geneva University Hospital
Locations (1):
- Geneva University Hospital/Division of Nephrology, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Triverio PA, Bridevaux PO, Roux-Lombard P, Niksic L, Rochat T, Martin PY, Saudan P, Janssens JP. Interferon-gamma release assays versus tuberculin skin testing for detection of latent tuberculosis in chronic haemodialysis patients. Nephrol Dial Transplant. 2009 Jun;24(6):1952-6. doi: 10.1093/ndt/gfn748. Epub 2009 Jan 22. PMID 19164327
- [Derived] Hadaya K, Bridevaux PO, Roux-Lombard P, Delort A, Saudan P, Martin PY, Janssens JP. Contribution of interferon-gamma release assays (IGRAs) to the diagnosis of latent tuberculosis infection after renal transplantation. Transplantation. 2013 Jun 27;95(12):1485-90. doi: 10.1097/TP.0b013e3182907073. PMID 23694948